CLINICAL TRIAL: NCT00668330
Title: Steroid Induced Osteoporosis in Patients With Systemic Lupus Erythematosus-Prevalence,Risk Factors and Treatment
Brief Title: Steroid Induced Osteoporosis in Patients With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SLE-2007-007
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Bone mineral density; ibandronate; alfacalcidol
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibandronate+alfacalcidol+calcium (Active Comparator): Bonviva
  Interventions: Drug: Ibandronate+alfacalcidol+calcium; Drug: placebo ibandronate+alfacalcidol+calcium
- Placebo ibandronate+alfacalcidol+calcium (Active Comparator)
  Interventions: Drug: Ibandronate+alfacalcidol+calcium; Drug: placebo ibandronate+alfacalcidol+calcium

INTERVENTIONS:
Drug: Ibandronate+alfacalcidol+calcium — Ibandronate 150 mg monthly plus daily alfacalcidol (1ug)500mg plus calcium
  Other Names: Bonviva
Drug: placebo ibandronate+alfacalcidol+calcium — placebo ibandronate monthly plus daily alfacalcidol(1ug)500mg calcium
  Other Names: placebo Bonviva

SUMMARY:
The primary aim of the present study was to investigate the prevalence of low bone mineral density (BMD) and vertebral fractures, as determined by a standardized assessment, and to elucidate the role of bone qualities, including micro-architecture, bone remodeling, bone turnover, mineralization and inflammation on bone density and prevalent vertebral fractures in a large population of systemic lupus erythematosus (SLE) patients.

The secondary aim of the study is to evaluate the following parameters in women with steroid induced OP (SIOP) before and after 1 year of treatment using:

1. The changes in BMD using dual energy X-ray absorptiometry (DXA)
2. Bone mineralization and architecture in-vivo using a newly available high-resolution human micro-computed tomography (ExtremCT), which can provide us with new insights into how the degree and distribution of mineralization are affected by long-term oral Ibandronate treatment.
3. Changes in perfusion and marrow edema before and after treatment of Ibandronate using dynamic Magnetic Resonance Imaging (MRI) in these patients with SIOP.
4. The investigators prospectively evaluate the correlation between the changes in brachial arterial endothelial function and lumbar spine BMD in female lupus patients over the period of 1 year.

DETAILED DESCRIPTION:
In the first part of the study, 150 consecutive patients with a diagnosis of SLE were included in the study. All patients fulfilled the American College of Rheumatology (ACR) revised criteria for the classification of SLE and provided written informed consent. Data collected at the time of study inclusion were age, disease duration, race, menstrual status, age at menopause, periods of amenorrhea, family history of osteoporosis, ultraviolet (UV) light intolerance, sunshine avoidance, use of sunscreens in the previous year, calculated mean daily dietary calcium intake in the last 3 months, history of (non)vertebral fractures after the age of 25 years, comorbidity, alcohol and tobacco intake, and exercise status.Body weight, height, and body mass index (BMI) were assessed. Disease activity was scored using the Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) 54. Accumulated organ damage was assessed with the SLICC/ ACR damage index (DI) 55. A modified DI score was derived as the DI score excluding osteoporotic fractures as a damage item.BMD measurements of the hip (total hip and femoral neck) and the lumbar spine (L1-4; anteroposterior view) as well as lateral radiographs of the thoracic and lumbar spine (T5-L4)were performed. The prevalence of low BMD and vertebral fractures will be assessed.

In the second part of the study, 40 female SLE patients with steroid induced osteopenia will be enrolled in a 12-month, randomized, parallel-group, controlled study. Patients will receive either oral Ibandronate 150 mg once monthly plus daily alfacalcidol (0.001 mg) or placebo ibandronate once monthly plus daily alfacalcidol(0.001mg).In addition, the intake of dietary calcium will estimate by a questionnaire on the screening visit. All patients will receive a daily calcium supplement(500 mg).

Primary outcome is the improvement of bone mineral density measured by DEXA.

Secondary outcome includes:

1. Evaluation of the changes in bone mineralization and architecture measured by Xtreme CT.
2. Evaluation of the changes in perfusion and marrow edema using MRI.
3. Anti-proliferative and anti-inflammatory action of alfacalcidol using serum level of interleukin-6 (IL-6), transforming growth factor-beta-1, angiotensin-II, as well as urinary levels of TGF and monocyte chemoattractant protein-1 (MCP-1).

ELIGIBILITY:
Part I

Inclusion Criteria:

* Fulfilled the ACR revised criteria for the classification of SLE
* Provided written informed consent for their participation

Part II

Inclusion Criteria:

* Have low BMD (T socre < -1 S.D. at the lumbar spine (L1-L4) or total hip) induced by the long-term administration of high-dose corticosteroids.
* Had been receiving chronic uninterrupted corticosteroid therapy for at least 1 year or had received a corticosteroid dose of at least 5 mg/day.

Exclusion Criteria:

* Hypocalcaemia, hypercalcaemia, Hypercalciuria, a creatinine clearance of less than 30 ml per minute.
* A history of nephrolithiasis during the previous five years.
* A history of recent major gastrointestinal (GI) tract disease (e.g. oesophagitis).
* Had or presence of primary hyperparathyroidism, hyperthyroidism, or hypothyroidism in the year before the study began.
* Had experienced any previous adverse reaction to bisphosphonate therapy (alendronate, fosamax, ibandronate).
* With uncontrolled active or recurrent peptic ulcer disease.
* Receiving therapy (within the last 6 months) known to affect bone metabolism, including:hormone-replacement agents, calcitonin, active vitamin D3 analogues, thiazide diuretics,treatment with bisphosphonates,fluoride treatment within the last 12 mons or for a total duration of 2 years; contraindications to calcium or vitamin D therapy.
* Pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome of Part I study is to investigate the prevalence of low BMD and vertebral fractures. Primary outcome of part II study is the improvement of bone mineral density measured by DEXA. | baseline and month 12

SECONDARY OUTCOMES:
Evaluation of the changes in bone mineralization and architecture measured by Xtreme CT. | baseline, month 6 and month 12
  The study will be analyzed using intention-to-treat (ITT) analysis
Evaluation of the changes in perfusion and marrow edema using MRI. | baseline, month 6, month 12
  The study will be analyzed using intention-to-treat (ITT) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- School of Pharmacy CUHK, Hong Kong, China

REFERENCES:
- [Derived] Li EK, Zhu TY, Hung VY, Kwok AW, Lee VW, Lee KK, Griffith JF, Li M, Wong KC, Leung PC, Qin L, Tam LS. Ibandronate increases cortical bone density in patients with systemic lupus erythematosus on long-term glucocorticoid. Arthritis Res Ther. 2010;12(5):R198. doi: 10.1186/ar3170. Epub 2010 Oct 22. PMID 20964867